14-03-2025

#### PATIENT INFORMATION SHEET

Before signing this informed consent form, please read the information below carefully and ask any questions you may have.

#### Nature:

The study aims to explore the use of biofrequency to assess nutritional markers using a noninvasive test, in addition to implementing a personalized nutritional intervention in a group of participants. Participation involves collecting a hair sample and completing questionnaires.

## Importance:

The research is innovative in its use of biofrequency, which could provide a faster, more accessible, and noninvasive method for assessing nutritional status, improving lifestyle habits, and preventing the onset of disease.

To conduct the study, a hair sample (3 strands) will be taken in a sterile, sanitary location. The protocol will last approximately 5 minutes, plus 20 minutes to complete a questionnaire (regarding nutritional and exercise habits, along with sociodemographic variables such as sex and age). All participants must be adults (18-65 years old).

The information donated for the study will be related to the biofrequencies determined by hair extraction, as well as the data provided in the questionnaire, which will be treated completely anonymously.

## Implications for the patient:

- Participation is entirely voluntary.
- The patient may withdraw from the study at any time, without giving any explanation and without this affecting his or her medical care.
- All personal data obtained in this study is confidential and will be processed in accordance with EU Regulation 2016/679 of the European Parliament and of the Council of April 27, 2016, on Data Protection (GDPR), and Organic Law 3/2018, of December 5, on the Protection of Personal Data and the Guarantee of Digital Rights. Therefore, it is important that you know the following information: In addition to the rights you already know (access, modification, objection, and deletion of data), you can now limit the processing of inaccurate data, request a copy, or request the transfer of the data you have provided for the study to a third party (portability). To exercise your rights, please contact the principal investigator of the study.
- The information obtained will be used exclusively for the specific purposes of this study.

### Risks of research for the patient:

No risks associated with participation are anticipated, as this is a non-invasive test. Data will be handled in accordance with data protection regulations, and participants may withdraw at any time.

If you require additional information, you can contact our studio staff at the following phone number: +34644170100 or by email: <a href="mailto:estudiocwba@gmail.com">estudiocwba@gmail.com</a>

You can also contact the Principal Investigator (David Manzano Sánchez, University of Almeria) at the following email address: dms700@ual.es

# **INFORMED CONSENT - WRITTEN CONSENT OF THE PATIENT**

# Application of a frequency measurement system for the measurement of nutritional biomarkers: Effects of a nutritional intervention on satisfaction and improvement of quality of life

I (First and Last Name):....

I have read the information document that accompanies this consent (Patient Information)

| • I was able to ask questions about the study "Application of a frequency measurement system measuring nutritional biomarkers: Effects of a nutritional intervention on satisfaction and improvem quality of life." | |
|---|---|
| I have received sufficient information about the study. I have spoken with the informing healt professional: | hcare |
| I understand that my participation is voluntary and I am free to participate or not in the study | <b>y</b> . |
| • I have been informed that all data obtained in this study will be confidential and will be trea accordance with Regulation (EU) 2016/679 of the European Parliament and of the Council of Ap 2016 on Data Protection (GDPR),Organic Law 3/2018, of December 5, on the Protection of Persona and the Guarantee of Digital Rights | ril 27 |
| • I have been informed that the donation/information obtained will only be used for the specific purposes of the study. | С |
| • I wish to be informed of my genetic and other personal data obtained during the course research, including any unexpected discoveries that may occur, provided that this information is nece to prevent serious harm to my health or that of my biological relatives. But | |
| I understand that I may withdraw from the study: | |
| <ul> <li>Whenever</li> <li>Without having to give explanations</li> <li>Without this affecting my medical care</li> </ul> | |
| • I freely agree to participate in the project entitled "Application of a frequency measurement sy for the measurement of nutritional biomarkers: Effects of a nutritional intervention on satisfaction improvement of quality of life." | |
| Patient's signatureProfessional's signature (or legal representative, if applicable) health informant | |
| Name and surname: | |